CLINICAL TRIAL: NCT00632242
Title: A Phase 2 Pilot Study of the Safety, Pharmacokinetics, and Pharmacodynamics of ARC1779 Injection in Patients With Von Willebrand Factor-Related Platelet Function Disorders
Brief Title: ARC1779 Injection in Patients With Von Willebrand Factor-Related Platelet Function Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Archemix Corp. (Industry)
Responsible Party: James Gilbert, MD, Chief Medical Officer, Archemix Corp.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARC1779-004
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2008-03

CONDITIONS: Purpura, Thrombotic Thrombocytopenic; Von Willebrand Disease Type-2b
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — ARC 1779

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- TTP Remission Cohort 1 (Experimental): Patients will receive a total dose of 0.47 mg/kg of ARC1779 over 4 hours to achieve a target plasma concentration of 6 mcg/mL
  Interventions: Drug: ARC1779
- TTP Remission Cohort 2 (Experimental): Patients will receive a total dose of 1.67 mg/kg of ARC1779 over 24 hours to achieve a target plasma concentration of 6 mcg/mL
  Interventions: Drug: ARC1779
- TTP Remission Cohort 3 (Experimental): Patients will receive a total dose of 3.34 mg/kg of ARC1779 over 24 hours to achieve a target plasma concentration of 12 mcg/mL
  Interventions: Drug: ARC1779
- Acute TTP Cohort 4 (Experimental): Patients will receive up to a total dose of 40.78 mg/kg of ARC1779 for ≤ 14 days to achieve a target plasma concentration of 12 mcg/mL
  Interventions: Drug: ARC1779
- vWD-Type2b Cohort 5 (Experimental): Subjects will receive either ARC1779, desmopressin or a combination of ARC1779 and desmopressin in a 3-period crossover design. The maximum dose of ARC1779 will be 0.47 mg/kg to achieve a target plasma concentration of 6 mcg/mL.
  Interventions: Drug: ARC1779

INTERVENTIONS:
Drug: ARC1779 — Initial stepwise infusion of 0.23 mg/kg given over 30 minutes and subsequent continuous infusion of an additional 0.24 mg/kg given over 4 hours at a rate of 0.001 mg/kg/min.
  Arms: TTP Remission Cohort 1
Drug: ARC1779 — Initial stepwise infusion of 0.23 mg/kg given over 30 minutes and subsequent continuous infusion of an additional 1.44 mg/kg given over 24 hours at a rate of 0.001 mg/kg/min.
  Arms: TTP Remission Cohort 2
Drug: ARC1779 — Initial stepwise infusion of 0.46 mg/kg over 30 minutes and subsequent continuous infusion of an additional 2.88 mg/kg given over 24 hours at a rate of 0.002 mg/kg/min.
  Arms: TTP Remission Cohort 3
Drug: ARC1779 — Initial stepwise infusion of 0.23 mg/kg given over 30 minutes and subsequent continuous infusion of an additional 1.44 mg/kg given over 24 hours at a rate of 0.001 mg/kg/min to produce a target plasma concentration of 6 mcg/mL.
  Continuous infusion of ARC1779 Injection may continue for ≤ 14 days. After initial 24 hours dose may be titrated to achieve a target plasma concentration of 12 mcg/mL as needed, on the basis of clinical and laboratory data, according to the Investigator's judgment.
  Arms: Acute TTP Cohort 4
Drug: ARC1779 — In one period of the sequence, ARC1779 will be administered to all subjects as a stepwise infusion of 0.23 mg/kg over 30 minutes and subsequent continuous infusion of an additional 0.24 mg/kg given over 4 hours at a rate of 0.001 mg/kg/min in combination with a dummy 30-minute infusion of placebo. In another period, subjects will receive a single infusion of desmopressin at a dose of 0.4 mcg/kg given over 30 minutes in combination with a dummy 30-minute stepwise infusion followed by 4-hour continuous infusion of placebo. In the one other period, subjects will receive the combination of desmopressin at a dose of 0.4 mcg/kg given over 30 minutes and ARC1779 given as a stepwise infusion of 0.23 mg/kg over 30 minutes and subsequent continuous infusion of an additional 0.24 mg/kg given over 4 hours at a rate of 0.001 mg/kg/min
  Arms: vWD-Type2b Cohort 5

SUMMARY:
To evaluate the overall safety and tolerability of ARC1779, a therapeutic oligonucleotide ("aptamer") in patients with three types of von Willebrand Factor related platelet disorders.

DETAILED DESCRIPTION:
ARC1779 Injection will be investigated in 4 cohorts of TTP patients as an uncontrolled, open-label study. Patients with vWD-2b will be enrolled in an additional cohort in a randomized, blinded, double-dummy, and placebo-controlled study.

Collectively, patients representing 3 different vWF-related platelet function disorders: TTP in remission, acute TTP, and vWD-2b will be treated in a total of 5 cohorts. Three cohorts will consist of patients who are status post an episode of TTP ("TTP Remission Cohorts") and will be treated with ARC1779 Injection in a dose- and duration-escalation design. In parallel, a single cohort of patients with acute TTP ("Acute TTP Cohort") will be treated according to an individual patient titration-to-response paradigm. This cohort will be opened for enrollment at the beginning of the study and closed after all of the other cohorts are completed. Also in parallel, a single cohort of patients with vWD-2b ("vWD-2b Cohort") will begin enrollment at the commencement of the study and continue independently of the course of the TTP Remission Cohorts. Up to 4 patients will be included in each of the TTP cohorts. The vWD-2b Cohort is expected to consist of up to 12 vWD-2b patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Age 18-75 years;
* vWD-2b - confirmed diagnosis, or;
* TTP Remission - prior episode(s) of primary acute TTP, or;
* Acute TTP - any episode, first or relapse, with presence of all of the following:

  1. Microangiopathic hemolytic anemia (schistocytosis present, Coombs test negative);
  2. Severe thrombocytopenia;
  3. Clinical diagnosis of either a primary or secondary form of TTP:(1) Primary TTP: e.g., familial TTP (Upshaw-Schulman syndrome), or acquired idiopathic TTP, or "atypical HUS"; (2) Secondary TTP: e.g., TTP occurring post-bone marrow transplant, drug-induced TTP, lupus-related TTP, etc.;
* Negative qualitative urine drug test at screening, and no history of alcohol or drug abuse;
* Not considering or scheduled to undergo any surgical procedure during the duration of the study;
* Has not donated or lost more than a unit of blood within 30 days prior to screening visit;
* Has not received an experimental drug within 30 days prior to screening;
* Female patients must be non-pregnant [for TTP Remission and vWD-2b Cohorts, a serum pregnancy test at screening and a urine pregnancy test at Day 1 pre-dose must be negative; for the Acute TTP Cohort, a serum pregnancy test at Day 1 pre-dose must be negative], and willing to use effective, redundant methods of contraception (i.e., for both self and male partner) throughout the study and for at least 30 days after participation. If possible, the treatment will be initiated within 5 days of the cessation of the preceding menstrual period;
* Male patients must agree to use a medically acceptable contraceptive (abstinence or use of a condom with spermicide) throughout the study and for at least 30 days after participation;
* Patients must be capable of understanding and complying with the protocol and must have signed the informed consent document prior to performance of any study-related procedures.

Exclusion Criteria:

* History of recent surgery or trauma;
* Any major, active health problem, e.g., cancer or heart disease, which could render the patient medically unstable during the period of participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To establish the overall safety and tolerability of ARC1779 in three varieties of von Willebrand Factor (vWF)-related platelet function disorders | 28 days

SECONDARY OUTCOMES:
To characterize the pharmacokinetic (PK) profile of ARC1779 intravenous (IV) infusion in patient groups | 28 days
To characterize the pharmacodynamic (PD) profile of ARC1779 in patients with vWF-related platelet function disorders with respect to parameters of platelet function and vWF activity | 28 days
To assess the concentration- and dose-response relationships among ARC1779 PK and PD parameters. | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Archemix Investigational Site, Vienna, Austria

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581